CLINICAL TRIAL: NCT02060994
Title: Respiratory Morbidity Among Children Who Were Born by Elective Cesarean Section After 37-38 Weeks vs. 39 Weeks and More
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Neonatologist, Hillel Yaffe Medical Center
Other Study IDs: HYMC-0088-13-CTIL
Record Dates: First submitted 2014-02-08; First posted 2014-02-12 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Respiratory Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 37-38 weeks: Children who were born by elective Cesarean section after 37-38 gestational weeks.
  Intervention: No intervention.
  Interventions: Other: No intervention
- 39 week or more: Children who were born by elective Cesarean section after 39 gestational weeks or more Intervention: No intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background: It is known that after Cesarean section is correlated with respiratory complication more, if done after 37-38 week of gestation than if done after 39 weeks or more.

Goal: The aim of the current study is to find out if these respiratory complications extend to later life.

Methode: Reviewing the patients' medical file, and collecting data about respiratory complication.

DETAILED DESCRIPTION:
Background: It is known that after Cesarean section is correlated with respiratory complication more, if done after 37-38 week of gestation than if done after 39 weeks or more. We have already conducted a study about this topic, and published our results.

Goal: The aim of the current study is to find out if these respiratory complications extend to later life.

Method: Reviewing the patients' medical file, and collecting data about respiratory complication. We will use the same patients we used at the first study. Respiratory complications are defined as diagnosis of asthma, treatment by inhalations or systemic steroids, or consultation by pulmonologist.

ELIGIBILITY:
Inclusion Criteria:

* Children born in 2007-2009 our medical center by elective Cesarean section according to a list of IDs we have.

Exclusion Criteria:

* Children with respiratory congenital defect that was not known at the first week of life.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born in 2007-2009 in "Hillel Yaffe" medical center by elective Cesarean section according to a list of IDs we have.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
There are respiratory complications. | Age 4-8 years
  Respiratory complications are defined as any of: asthma, inhalation therapy, systemic steroids therapy, consultation by a pulmonologist

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillle Yaffe medical center, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, North, Israel

REFERENCES:
- [Background] Nir V, Nadir E, Feldman M. Late better than early elective term Cesarean section. Acta Paediatr. 2012 Oct;101(10):1054-7. doi: 10.1111/j.1651-2227.2012.02772.x. Epub 2012 Jul 16. PMID 22758608